CLINICAL TRIAL: NCT07194603
Title: Association Between Conditioned Pain Modulation and the Longitudinal Response to Spinal Mobilization in Adults With Chronic Neck Pain
Brief Title: Association Between Conditioned Pain Modulation and the 4-week Response to Spinal Mobilization in Adults With Chronic Neck Pain
Acronym: CPMNeck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azusa Pacific University (Other)
Collaborators: Sacred Heart University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-141; T42OH008422 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain Musculoskeletal; Chronic
Keywords: conditioned pain modulation; joint mobilization; spinal mobilization; chronic neck pain; pain pressure threshold; cold pressor test; numeric pain rating scale; neck disability index; global perceived recovery
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: It is a cohort intervention study
Masking Description: Everyone, including the outcome assessor, was blinded to what the conditioned pain modulation was for each participant throughout the data collection session. The researcher applying the algometer for the pain pressure threshold did not record the values, instead the outcomes assessor did this step. Although the outcome assessor recorded the pain pressure thresholds (PPTs) pre-/post-cold pressor test [PPTs are used to calculate the conditioned pain modulation before AND after the intervention], they did not calculate the conditioned pain modulation until the end of the data collection day when all the participants have left.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal/joint mobilization of the neck (Experimental): The principal investigator provided spinal mobilization (SM) of the neck consisting of grade III unilateral postero-anterior (PA) and antero-posterior (AP) oscillatory joint mobilization (JM) to the cervical spine [5 minutes of PA and 5 minutes of AP in random order based on the random sequence for the CPM measurement] for a total of 10 minutes to the patient's most painful cervical spine segment/s. Both SM and JM mean the same thing and are synonymous. Prior to SM, the PI explained why SM might work and advised participants to continue their usual activities of daily living.
  Interventions: Procedure: Spinal mobilization (SM) of the neck

INTERVENTIONS:
Procedure: Spinal mobilization (SM) of the neck — This cohort intervention study has only one arm and this arm has only one intervention, the one described above. Both SM and JM mean the same thing and are synonymous.

SUMMARY:
The goal of this observational study is to learn if there is a relationship between conditioned pain modulation or CPM (a test of your brain's ability to inhibit pain) and longitudinal clinical outcomes following one spinal/joint mobilization (commonly used to treat neck pain) session in individuals with chronic mild neck pain between the age of 18-55 years old. The main questions it aims to answer are:

* Is baseline CPM significantly associated with baseline outcomes: (a) pain (NPRS), (b) perceived disability (NDI), and (c) perceived recovery (GPR)?
* Is baseline CPM associated with longitudinal trend in outcomes: pain (NPRS), perceived disability (NDI), and perceived recovery (GPR)?
* Is the change in CPM post-joint mobilization (post-JM) associated with longitudinal trend in outcomes: pain (NPRS), perceived disability (NDI), and perceived recovery (GPR)? Participants will receive CPM protocol before and after the joint mobilization. The CPM protocol includes a handheld pressure meter applied to 3 main sites (neck, shoulder blade and leg bone) to measure when light touch first becomes a mild experience of pain as well as placing your hand in cold water. They will receive joint/spinal mobilization of the neck (cervical spine), explanation of why it might work and advise to continue their usual activities of daily living and to avoid receiving any physical therapy treatments/interventions (such as exercise or joint mobilization; they may continue taking their medication/s, however) the entire 4-weeks while they are in the study.

DETAILED DESCRIPTION:
It has been proposed that neck joint mobilization (JM) [also known as spinal mobilization (SM) of the neck] reduces pain by targeting conditioned pain modulation (CPM) Two studies support the theory that pain relief from JM is the result of processing occurring in the brainstem, the region where CPM is housed. A study found that one exposure of JM normalized impaired CPM and reduced pain. Another study suggested that CPM and JM may share a common CNS pathway from the brainstem to the spinal cord. If so, this may explain the mechanism by which JM relieves pain. Understanding these relationships may allow clinicians to better target treatment to those who may benefit from a JM intervention, potentially reducing the burden associated with chronic neck pain. The purpose of this study is to explore the relationship between CPM and clinical outcomes following JM in those with mild chronic neck pain. This is the first study investigating these relationships.

SPECIFIC AIMS Aim 1: To determine the impact of one JM treatment on CPM and clinical outcomes in patients with chronic neck pain and associated disorder type I (NAD I) or mild neck pain.

Aim 2: To explore these relationships longitudinally. HYPOTHESES [Primary hypotheses]

1. Baseline CPM is significantly associated with baseline outcomes: (a) pain (Numeric pain rating scale or NPRS), (b) perceived disability (Neck disability index or NDI), and (c) perceived recovery (global perceived recovery or GPR).
2. Baseline CPM is associated with longitudinal trend in outcomes: pain (NPRS), perceived disability (NDI), and perceived recovery (GPR)
3. Change in CPM post-JM is associated with longitudinal trend in outcomes: pain (NPRS), perceived disability (NDI), and perceived recovery (GPR)

RESEARCH QUESTIONS

1. What is the baseline CPM in a community sample of individuals with chronic mild neck pain (CNP)?
2. What is the prevalence of impaired CPM at baseline in a community sample of individuals with CNP?
3. In the subgroup of CNP with impaired baseline CPM readings, what proportion has normalized CPM readings, immediately following JM?

EXPERIMENTAL DESIGN AND METHODS Study design. A prospective, longitudinal, cohort study with intervention Sample size. 31 participants were enrolled. Subject recruitment. Participants were recruited via (1) emails sent to the Sacred Heart University (SHU) and Azusa Pacific University community; (2) flyers posted in physical therapy clinics within 30 miles of SHU, and (3) social media advertisements. All recruitment materials specified the study details. Potential subjects who responded were screened by research assistants over the phone, via email, or via a QR coded questionnaire embedded in the flyer to determine eligibility based on the inclusion and exclusion criteria. Patients who met the inclusion criteria were invited to meet with the research assistants, who explained the study and obtained informed consent. Eligible participants were instructed to wear non-restrictive clothing and to refrain from taking analgesics, serotonin norepinephrine reuptake inhibitors (SNRIs), and opioids for 24 hours before CPM data collection.

Venue. Sacred Heart University and Azusa Pacific University physical therapy departments Demographic and clinical variables. Demographic and clinical variables were collected, including age, sex, body mass index (BMI) (calculated based on weight and height), and pain medications (analgesics, SNRIs, opioids). A critical factor in determining the success or failure of conservative care is healthcare utilization (pre- and post-JM). The total number of visits during the study period was tabulated.

Procedure/Methods. The principal investigator (PI) trained assistants/associates to facilitate PI blinding. Patients who consented were assessed for baseline CPM, NDI, and NPRS.

The PI has been practicing orthopedic physical therapy for more than 20 years. He is a manual therapy fellowship-trained and board-certified orthopedic physical therapy clinical specialist. Prior to the baseline CPM assessment, the assistant took the blood pressure and heart rate of the subject, and the investigator conducted a clinical examination assessing the active range of motion and a manual examination to identify the most painful segmental level using both the unilateral postero-anterior (PA) and antero-posterior (AP) oscillatory JM techniques and to familiarize the patient with these two JM techniques which were performed as intervention. Following baseline CPM assessment, there was a 15-minute rest period when the PI provided information on the natural history of neck pain, how JM is believed to work, and the ability to fully participate in usual activities after treatment. Patients were also told to avoid other JM or exercise treatments during the 4-week follow-up period. Next, the PI provided grade III unilateral PA and AP oscillatory JM (5 minutes of PA and 5 minutes of AP in random order based on the random sequence for the CPM measurement such that #1 is for PA and #2 or #3 is for AP) for a total of 10 minutes to the patient's most painful cervical spine segment/s. This dose of JM is based on the work of a study whose authors demonstrated improved pain and global perceived effect. Immediately following JM, research team member #2 reassessed CPM (called post-JM CPM) and later subtracted it from the baseline CPM reading. This is hereby referred to as "change in CPM." After the associate investigator measured post-JM CPM, the participant's blood pressure and heart rate were measured a second time as JM has been shown to affect these vital signs. The purpose was to ensure that was no adverse cardiovascular response to the intervention. At 2 days, 2-, and 4-weeks following JM, a research team associate made a follow-up phone call, sent a text reminder, and/or email request to examine the NPRS score, NDI, GPR, and other clinical variables (e.g., pain medication use, number of healthcare visits related to neck pain). Participants were reminded to avoid receiving JM or exercise interventions for the 4 weeks study period.

To maintain the fidelity of the intervention and protocol, another professor of orthopedic physical therapy (who taught JM for more than 5 years) randomly observed the data collection processes and treatment administration.

Statistical analysis. The characteristics of subjects, including demographics and baseline clinical measurements, were summarized using descriptive statistics, the median, and interquartile range for continuous variables (e.g., age, CPM, NPRS, GPR, NDI, and BMI) and percentages (counts) for categorical variables (ex. sex). All statistical tests were two-sided, and a value of p<0.05 was considered statistically significant. All continuous outcome variables were checked for normality using the Shapiro-Wilk test prior to the statistical analyses.

For hypotheses 1 a linear regression model was used to evaluate the potential association between baseline CPM and three dependent variables (NPRS, NDI, GPR) in a univariate manner and then a multivariate linear regression manner.

For hypotheses 2 and 3, a linear mixed-effect regression (MEM) model was used to evaluate whether baseline CPM or a change in CPM (respectively) is associated with a longitudinal trend in change in pain, GPR, or function (NDI) with baseline as the reference, at 2-day, 2 week, and 4 week follow up adjusting for patient baseline demographics (age, sex, and BMI). The MEM was specified with random intercepts and slopes such that a linear trajectory representing outcome values was compared. Individual-level specific intercept and slopes over the period of follow-up were included as random effects, while other covariates were modelled as fixed effects. All models were adjusted for other baseline clinical (including CPM) and demographic confounders. Residual-based diagnostics were used to evaluate the validity of model assumptions. Secondarily, to test hypotheses 2 and 3 for single time points, linear regression analyses were performed with univariate analyses conducted first, and if the cutoff p-value of 0.10 was met for a variable, then the multivariate analysis followed. Once included in the multivariate model, a p-value of < 0.05 was considered significant.

For research question #1, descriptive statistics were used to answer the question regarding the baseline CPM levels in the study sample. Research questions #2 and #3 were answered by examining the proportions of participants with impaired CPM at baseline and from this subgroup, determining how many have normalized CPM post-JM.

ELIGIBILITY:
Inclusion Criteria:

* neck pain classified as Neck Pain and Associated Disorder I (NAD) I with a duration of 3-60 months
* a 3 or higher pain scale rating out of 10 on the Numeric Pain Rating Scale
* modified STarTBack tool (modified for neck pain) classified as low risk (< 3 out of 9)
* a Neck Disability Index scored at 10% or higher

Exclusion Criteria:

* prior spinal surgery, those with serious underlying pathology including neurologic, cardiovascular, hypertension, diabetes mellitus, inflammatory arthritis, osteoporosis, hemophilia, cancer, contra-indications to cervical spine joint mobilization (or spinal mobilization of the neck) [e.g., a history of fainting spells or loss of consciousness, presently on blood thinners]
* those who received spinal mobilization of the neck (or cervical spine joint mobilization) or physical therapy prescribed exercise in the past 3 months, current smokers, those with chronic widespread pain, those actively pursuing compensation, unable to work or with litigation pending or unable to communicate in English, persons who cannot tolerate 2 minutes of the cold pressor test (12 degrees Centigrade).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | NPRS was taken at baseline- on the day of the data collection and prior to receiving the intervention. Follow-up NPRS were collected at: 2 days, 2 weeks and 4 weeks after baseline (baseline= is the date receiving the intervention)
  The NPRS is a self-reported measure of the intensity of pain from 0 (no pain) to 10 (worst possible pain). It can be reported verbally (and has been validated for reporting by telephone), administered graphically on screen or on paper.
Baseline Conditioned Pain Modulation | Before spinal/joint mobilization of the neck or cervical spine
  Measuring CPM involves three steps. In step one (test stimulus) a pressure algometer is applied randomly to 3 marked anatomical sites (i.e., symptomatic side of the neck at C3/4, infraspinatus of the shoulder and the anterior tibial muscle of the lower extremity to determine the pain pressure threshold or PPT). The pressure is applied to the patient until the pressure is first perceived as pain, and the pressure value is recorded.
  Step two (conditioning stimulus) is the cold pressor test or CPT, which involves placing the hand in a basin of cold water (12 degrees Centigrade) for 2 minutes.
  Step three (test stimulus) is a repeat of step one. CPM= [PPT (step 3) minus PPT (step 1)] divided by PPT (step 1) * 100. The CPM is expressed as a %.
  CPM= (PPT (step 3)-PPT (step 1))/(PPT (step 1)) × 100 A positive number signifies a normal CPM. No change or a negative number indicates an abnormal CPM.
Change in CPM (change in conditioned pain modulation) | Immediately after the intervention (spinal mobilization)
  Change in CPM: is the difference between post-intervention (post-JM) CPM and baseline CPM. Post-JM CPM is assessed after spinal/joint mobilization of the neck or cervical spine using the same procedure as when the baseline CPM was assessed. Thus, Post-JM CPM minus baseline CPM= Change in CPM. How CPM is measured is described under "baseline CPM" above.

SECONDARY OUTCOMES:
Global perceived recovery (GPR) | GPR was taken at baseline- on the day of data collection and prior to receiving the intervention to determine patient expectation of recovery at 4-weeks. Follow-up GPR were collected at: 2 days, 2 weeks and 4 weeks after the date of the intervention.
  Global perceived recovery (GPR), an indicator of overall perceived recovery, is an important discharge criterion that can be utilized in physical therapy practice and is measured by asking "how well do you feel you are recovering from your injuries?" The response options are: (1) completely better, (2) much improved, (3) slightly improved, (4) no change, (5) slightly worse, (6) much worse, (7) worse than ever. Response options (1) and (2) signify that the participants have met the discharge criterion when used in the clinical setting.
Neck Disability Index (NDI) | NDI was taken at baseline- on the day of the data collection prior to receiving the intervention. Follow-up NDI were collected at: 2 days, 2 weeks and 4 weeks after baseline (baseline= the date receiving the intervention)
  The NDI is a self-report of cervical spine or neck function from 0-100%, 0% indicates no disability and higher values indicate more severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Yung, PT, DPT, Principal Investigator — New York University (at the time of the study)
Locations (1):
- Azusa Pacific University, Azusa, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data set which includes all outcome measures described in the study will be shared upon publication of this original study in an indexed peer-reviewed journal once it is available in print.
Supporting Information: Study Protocol, SAP
Time Frame: Start date: Upon publication of the original study in an indexed peer-reviewed journal once it is available in print. End date: one year from the start date
Access Criteria: Anyone can access this data set.
URL: https://figshare.com/